CLINICAL TRIAL: NCT03421483
Title: Factors Affecting Colonic Folate Absorption and Metabolism in Humans
Brief Title: Assessing Colonic Folate Absorption & Metabolism
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Natural Sciences and Engineering Research Council, Canada (Other)
Responsible Party: Principal Investigator, Deborah O'Connor, Senior Associate Scientist, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 1000059584
Record Dates: First submitted 2018-01-08; First posted 2018-02-05 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Folate
Keywords: Folate; Absorption; Metabolism; Colon; Receptor; Enzyme

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Folic Acid supplementation (Active Comparator): Participants receive an adult multivitamin supplement along with a folic acid supplement
  Interventions: Dietary Supplement: Folic Acid supplementation; Dietary Supplement: Adult Multivitamin
- No supplementation (Placebo Comparator): Participants only receive an adult multivitamin supplement
  Interventions: Dietary Supplement: Adult Multivitamin

INTERVENTIONS:
Dietary Supplement: Folic Acid supplementation — Participants receive a 400 microgram Folic Acid supplement
  Arms: Folic Acid supplementation
Dietary Supplement: Adult Multivitamin — Participants will receive an adult multivitamin supplement

SUMMARY:
Folate, a B-vitamin, is necessary in metabolic processes such as amino acid and nucleotide synthesis. Since folate cannot be synthesized by mammals, it must be consumed as foods and dietary supplements or generated by bacteria present in the colon. There are many known adverse health outcomes associated with folate deficiency in humans such as neural tube defects in newborns and colorectal cancer in adults. It has also been proposed that supra-physiological folate status can also be detrimental since it can lead to changes in immune function and the masking of vitamin B12 deficiency. It is generally believed that dietary sources of folate are primarily absorbed in the small intestine, however recent evidence suggests the colon may play a more significant role in the absorption of folate than previously understood. The aim of this study is to assess how folic acid supplementation influences colonic folate absorption and metabolism in humans. This will be accomplished by assessing the expression of two major folate transporters responsible for folate absorption in the colon. Participants will be randomized to receive multivitamins with either 0 or 400 µg folic acid during a 16-week randomized clinical trial in which blood and colonic tissue biopsies will be collected and analyzed. The total folate concentrations and expression of folate transporters in colonocytes will be measured to confirm levels and evaluate the impact of supplemental folic acid. The expression of two folate hydrolases responsible for converting naturally occurring folate to its bioavailable form will also be evaluated. This work will lead to a deeper understanding of colonic folate absorption and metabolism, resulting in more appropriate dietary and supplemental folate recommendations.

DETAILED DESCRIPTION:
The vitamin folate is necessary for one-carbon metabolism in processes such as amino acid and nucleotide synthesis. As folate cannot be synthesized by mammals, it must be sourced from the diet and dietary supplements or generated by bacterial species present in the colon. There are a number of well-established adverse health outcomes associated with folate deficiency in humans, including congenital neural tube defects in newborns and colorectal cancer in adults. It has been proposed supra-physiological folate status can also be detrimental since it can lead to changes in immune function and the masking of vitamin B12 deficiency. It is generally believed that dietary sources of folate are primarily absorbed in the small intestine, however recent evidence from our team and others suggests that the colon may play a greater role in absorption of folate than previously understood. Specifically the amount of folate in the colon, much of it generated by the microbiome, can exceed dietary intakes of folate from natural sources. There are a number of gaps in knowledge regarding colonic folate absorption in humans. It is not known to what degree folate specific transporters such as proton coupled folate transporter (PCFT) and reduced folate carrier (RFC) are present in the colon of healthy humans. To date, the majority of studies conducted identifying the presence of RFC and PCFT in colonocytes have been performed using cell lines or tissue harvested from organ donors. To our knowledge, no study has investigated the mRNA and protein concentrations of both RFC and PCFT present in human colonic tissue retrieved as biopsies. It also remains to be determined if folate status influences RFC and PCFT expression at the level of the colon. Secondly, it remains unclear to what degree the two intestinal folate hydrolases, glutamate carboxypeptidase II (GCPII) and γ-glutamyl hydrolase (GGH) are present in colonic mucosa. To gain a more thorough understanding of the fundamental processes involved in folate absorption in the colon of humans, the following three objectives are proposed. The primary objective is to evaluate the impact of 0 and 400 µg supplemental folic acid on total folate concentrations within the colonic mucosa by measuring folate levels. The secondary objectives include evaluating the impact of 0 and 400 µg supplemental folic acid on the regulation of PCFT and RFC in the ileum and colon by assessing the expression of mRNA transcripts and proteins, and determining the degree to which GCPII and GGH are present in the lumen of the ileum and colon by quantifying enzyme activity and expression of mRNA transcripts and proteins. To accomplish this, a 16-week longitudinal open-labelled randomized clinical trial will be conducted. Recruitment and screening will require three separate steps comprised of an initial invitation to participate, followed by a telephone screening session to determine eligibility and finally a baseline in-person study visit prior to enrollment into the intervention phase of the study. Once enrolled, participants will be asked to follow a diet low in synthetic folic acid for the duration of the study. At enrollment, subjects will be randomized to receive a multivitamin supplement and either 0 or 400 µg folic acid. Follow-up study visits will take place at week 8 and week 16 where anthropometric measurements, blood and colonic tissue biopsies (Week 16 only) from the terminal ileum, cecum, ascending colon, and descending colon will be collected for analysis. 24-hour dietary recalls will be collected throughout the study to observe folate and caloric intake. Plasma, RBC folate levels, and colonic mucosa folate content will be determined via microbial assay. GCPII and GGH enzyme activity will be determined according to the Krumdieck and Baugh method with modification. PCFT and RFC expression will be determined via semi-quantitative real-time PCR and protein samples will be extracted in a Western Blot Analysis using RIPA lysis and extraction buffer. The proposed study will further our understanding of the fundamental processes of folate metabolism and absorption in the colon. Results from this study may help to establish the optimal intakes of dietary folate, meeting the requirements of humans, without the potential health risks related to over-exposure to folate.

ELIGIBILITY:
Inclusion Criteria:

1. Males >18 years old and <75 years old;
2. Females who are pre-menopausal that have had a hysterectomy or tubal ligation, post-menopausal (at least 1 year) and <75 years old;
3. Describe themselves as generally healthy.
4. Recommended to have a colonoscopy examination by their Doctor

Exclusion Criteria:

1. They have a history of gastrointestinal disease (such as Crohn's disease, ulcerative colitis, celiac disease) and/ or gastrointestinal cancers;
2. They have had a previous colon resection;
3. They are regularly using medications that may affect gastrointestinal pH or folate metabolism (e.g. proton pump inhibitors, phenytoin, phenobarbital, primidone, or have used oral antibiotics within the last 2 weeks);
4. On a regular basis they consume >2 alcoholic drinks/day for women or >3/day for men;
5. They are currently smokers;
6. They are folic acid supplement users or have used folic acid supplements or multivitamins containing folic acid in the last 4 months;
7. They have a bleeding disorder (such as hemophilia)
8. They are unlikely able to discontinue anti-coagulant therapy prior to colonoscopy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2018-12-17 (Actual); Primary Completion 2023-10-15 (Estimated); Study Completion 2023-10-15 (Estimated)

PRIMARY OUTCOMES:
Colonic folate levels | 4 months
  Evaluate the impact of 0 and 400 µg supplemental folic acid on total folate concentrations within the colonic mucosa by measuring folate levels

SECONDARY OUTCOMES:
PCFT | 4 months
  Evaluate the impact of 0 and 400 µg supplemental folic acid on the regulation of PCFT in the ileum and colon by assessing the expression of mRNA transcripts and proteins
RFC | 4 months
  Evaluate the impact of 0 and 400 µg supplemental folic acid on the regulation of RFC in the ileum and colon by assessing the expression of mRNA transcripts and proteins
GCPII | 4 months
  Determine the degree to which GCPII is present in the lumen of the ileum and colon by quantifying enzyme activity and expression of mRNA transcripts and proteins
GGH | 4 months
  Determine the degree to which GGH is present in the lumen of the ileum and colon by quantifying enzyme activity and expression of mRNA transcripts and proteins

CONTACTS AND LOCATIONS:
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Institute of Medicine (US) Standing Committee on the Scientific Evaluation of Dietary Reference Intakes and its Panel on Folate, Other B Vitamins, and Choline. Dietary Reference Intakes for Thiamin, Riboflavin, Niacin, Vitamin B6, Folate, Vitamin B12, Pantothenic Acid, Biotin, and Choline. Washington (DC): National Academies Press (US); 1998. Available from http://www.ncbi.nlm.nih.gov/books/NBK114310/ PMID 23193625
- [Background] Said HM. Intestinal absorption of water-soluble vitamins in health and disease. Biochem J. 2011 Aug 1;437(3):357-72. doi: 10.1042/BJ20110326. PMID 21749321
- [Background] Mason JB, Tang SY. Folate status and colorectal cancer risk: A 2016 update. Mol Aspects Med. 2017 Feb;53:73-79. doi: 10.1016/j.mam.2016.11.010. Epub 2016 Nov 24. PMID 27890600
- [Background] De Wals P, Tairou F, Van Allen MI, Uh SH, Lowry RB, Sibbald B, Evans JA, Van den Hof MC, Zimmer P, Crowley M, Fernandez B, Lee NS, Niyonsenga T. Reduction in neural-tube defects after folic acid fortification in Canada. N Engl J Med. 2007 Jul 12;357(2):135-42. doi: 10.1056/NEJMoa067103. PMID 17625125
- [Background] Lakoff A, Fazili Z, Aufreiter S, Pfeiffer CM, Connolly B, Gregory JF 3rd, Pencharz PB, O'Connor DL. Folate is absorbed across the human colon: evidence by using enteric-coated caplets containing 13C-labeled [6S]-5-formyltetrahydrofolate. Am J Clin Nutr. 2014 Nov;100(5):1278-86. doi: 10.3945/ajcn.114.091785. Epub 2014 Sep 3. PMID 25332326
- [Background] Qiu A, Jansen M, Sakaris A, Min SH, Chattopadhyay S, Tsai E, Sandoval C, Zhao R, Akabas MH, Goldman ID. Identification of an intestinal folate transporter and the molecular basis for hereditary folate malabsorption. Cell. 2006 Dec 1;127(5):917-28. doi: 10.1016/j.cell.2006.09.041. PMID 17129779
- [Background] Dudeja PK, Torania SA, Said HM. Evidence for the existence of a carrier-mediated folate uptake mechanism in human colonic luminal membranes. Am J Physiol. 1997 Jun;272(6 Pt 1):G1408-15. doi: 10.1152/ajpgi.1997.272.6.G1408. PMID 9227476
- [Background] Kumar CK, Moyer MP, Dudeja PK, Said HM. A protein-tyrosine kinase-regulated, pH-dependent, carrier-mediated uptake system for folate in human normal colonic epithelial cell line NCM460. J Biol Chem. 1997 Mar 7;272(10):6226-31. doi: 10.1074/jbc.272.10.6226. PMID 9045638
- [Background] Paniz C, Bertinato JF, Lucena MR, De Carli E, Amorim PMDS, Gomes GW, Palchetti CZ, Figueiredo MS, Pfeiffer CM, Fazili Z, Green R, Guerra-Shinohara EM. A Daily Dose of 5 mg Folic Acid for 90 Days Is Associated with Increased Serum Unmetabolized Folic Acid and Reduced Natural Killer Cell Cytotoxicity in Healthy Brazilian Adults. J Nutr. 2017 Sep;147(9):1677-1685. doi: 10.3945/jn.117.247445. Epub 2017 Jul 19. PMID 28724658
- [Background] Chakraborty H, Nyarko KA, Goco N, Moore J, Moretti-Ferreira D, Murray JC, Wehby GL. Folic Acid Fortification and Women's Folate Levels in Selected Communities in Brazil - A First Look. Int J Vitam Nutr Res. 2014;84(5-6):286-94. doi: 10.1024/0300-9831/a000215. PMID 26255550
- [Derived] Farrell CC, Khanna S, Hoque MT, Plaga A, Basset N, Syed I, Biouss G, Aufreiter S, Marcon N, Bendayan R, Kim YI, O'Connor DL. Low-dose daily folic acid (400 mug) supplementation does not affect regulation of folate transporters found present throughout the terminal ileum and colon of humans: a randomized clinical trial. Am J Clin Nutr. 2024 Mar;119(3):809-820. doi: 10.1016/j.ajcnut.2023.12.018. Epub 2023 Dec 28. PMID 38157986